CLINICAL TRIAL: NCT03083756
Title: Prospective Observational Study for the Validation of a Risk Score Opportunistic Infections Development in Kidney Transplant Patients
Brief Title: Validation of a Risk Score Opportunistic Infections Development in Kidney Transplant Patients
Acronym: SIMPLICITY
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Trasplante (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: SET-INF-2014-01
Record Dates: First submitted 2017-03-08; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Opportunistic Infections
MeSH Terms: conditions — Opportunistic Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study validate the usefulness of SIMPLICITY score to characterize the immune status of the kidney transplant receiver at two points along its course (the one and six months after transplantation), by determination in peripheral blood of various parameters related to cellular immunity (count subpopulations of CD3+ (cluster of differentiation 3), CD4+ (cluster of differentiation 4) and CD8+( cluster of differentiation 8)), humoral immunity (immunoglobulins count) and innate (complement).

DETAILED DESCRIPTION:
The monitoring of various parameters related to cellular and humoral immunity (lymphocytes, immunoglobulins and complement) through a score (SIMPLICITY) (8) would allow the identification of renal transplant recipients at high risk for post-transplant infection. Prolonged or prolonged use of CMV (Cytomegalovirus) prophylaxis may modify this risk.

The SIMPLICITY score (Seeking for Immune Status based on Peripheral Blood Lymphocytes, Immunoglobulins and Complement Activity) is a practical score based on the monitoring of readily available immunological parameters to assess the risk of infection after RT (Renal transplant). In order to perform this score, the total lymphocyte counts and peripheral blood lymphocyte subpopulations (PBLSs), serum immunoglobulin levels (IgG, IgA (Immunoglobulin A) and IgM) and serum complement levels (C3 and C4) at baseline were investigated, at one month and 6 months after transplantation.

The validation of this new score would allow to have a weapon that would lead to reduce to the maximum the pharmacological immunosuppression and to use strict prophylactic measures in these patients.

The results of the present study may provide insight into clinically and scientifically relevant aspects of infection in the recipient of an RT undergoing immunosuppressive therapy:

From the point of view of assistance, if the hypothesis of the study were confirmed, the possibility of elaborating specific strategies of prophylaxis and early treatment (antibiotic, antifungal or antiviral), adjusted to the risk of the recipient to present some infectious event during its evolution post transplantation according to the SIMPLICITY score.

Likewise, it could lay the foundations for the design of individualized immunosuppression guidelines, in which the risk of infectious complications could be evaluated jointly with that of graft rejection. And all this based on simple immunological parameters, of economic determination and accessible for most of the centers of our environment, circumstance that would favor its immediate application in the usual clinical practice.

Given that the literature on this line of research is scarce, and the hypothesis we intend to demonstrate is novel and conceptually attractive, the results of this study will be able to be published in journals with a high impact index in the field of immunology and Management of infectious complications in the RT.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patients whose variables can be properly monitored throughout the first year post-transplant.
* Older than 18 years.
* Patients who have signed the informed consent form.

Exclusion Criteria:

* Infection with the human immunodeficiency virus (HIV).
* Patient who dies during the first month after transplant.
* Pre-transplant diagnosis of primary immunodeficiency (eg. Common variable immunodeficiency, idiopathic CD4 lymphopenia, etc)
* Patient is participating in another clinical trial with a molecule under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2014-08; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
To validate SIMPLICITY Score to characterize the immunological situation of the RT recipient at month of transplantation). | At 1 month from transplant
  To validate the SIMPLICITY will be scored from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD8+ (<0.200x103/MicroL at month 1)
To validate SIMPLICITY Score to characterize the immunological situation of the RT recipient at six months of transplantation. | At 6 months from transplant
  To validate the SIMPLICITY will be scored from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD3+ (<0.500x103 MicroL at 6 months).

SECONDARY OUTCOMES:
Correlation of IgG and infectious complications | Up to 12 moths from transplant
  Correlation of IgG and the incidence of infectious complications increased.
Correlation of C3 and infectious complications | Up to 12 moths from transplant
  Correlation of C3 and the incidence of infectious complications increased.
Correlation of count lymphocyte T CD3+ in Peripheral blood and infectious complications | Up to 12 moths from transplant
  Correlation count of lymphocyte subpopulations CD3+ and the incidence of infectious complications increased.
Correlation of count lymphocyte T CD8+ in Peripheral blood and infectious complications | Up to 12 moths from transplant
  Correlation count of lymphocyte subpopulations CD8+ and the incidence of infectious complications increased.
Acute rejection with histologic confirmation by conventional criteria | Up to 12 moths from transplant
  Number of patients who have had at least one acute biopsy-proven rejection throughout the study.
Graft loss with or without retransplantation. | Up to 12 moths from transplant
  Number of patients who have lost the graft throughout the study.
Mortality infectious cause | Up to 12 moths from transplant
  Number of dead patients and whose cause of death is Infection.
Mortality otherwise. | Up to 12 moths from transplant
  Number of dead patients whose cause of death has indicated a different cause to Infection (ie the reason for death was due to ischemic heart disease, or by another cardiovascular complication, or by neoplastic disease or by others).
CMV infection/Disease | Up to 12 moths from transplant
  Percentage of patients presenting at least one CMV disease throughout the study, from the transplant and number of CMV diseases per patient.
CMV viremia | Up to 12 moths from transplant
  Number of patients who had CMV positive viremia (either PCR (Polymerase Chain Reaction) or antigenemia) at least during one visit (No. of copies>0 IU/mL in PCR or>100,000/cell in Antigenemia).
To analyze the influence of low lymphocyte count in the increase of the rate of major infectious complications. | Up to 12 moths from transplant
  Low lymphocyte count, defined as lymphocytes <1500 cells/mcl and the rate of major infectious complications
To analyze the influence of CMV serology in the increase of the rate of major infectious complications. | Up to 12 moths from transplant
  CMV receptor serology vs. donor CMV Serology (ie, a new categorical variable will be constructed combining donor and recipient serology: D+/R+, D-/R +,D-/R-, D+/R-) and the rate of major infectious complications
To analyze the influence of Historical PRA (Panel Reactive Antibody) in the increase of the rate of major infectious complications | Up to 12 moths from transplant
  Historical PRA (%) and the rate of major infectious complications
To analyze whether viremia has any impact on the occurrence of other opportunistic diseases | Up to 12 moths from transplant
  Presence of major post-transplant infectious complication and the occurrence of other opportunistic diseases.
To analyze whether CMV disease has any impact on the occurrence of other opportunistic diseases. | Up to 12 moths from transplant
  Presence of CMV disease and the occurrence of other opportunistic diseases.
To analyze the role of Anticipated treatment and the influence in the appearance of infection or disease by CMV. | Up to 12 moths from transplant
  Indication of Anticipated treatment and appearance of infection or disease by CMV.
To analyze the role of Antiviral prophylaxis and the influence in the appearance of infection or disease by CMV. | Up to 12 moths from transplant
  Indication of Antiviral prophylaxis appearance of infection or disease by CMV.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 1 month of transplantation on overall survival throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 1 month of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD8+ (<0.200x103/MicroL at month 1)) and overall survival throughout the first year of evolution.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 1 month of transplantation on graft survival throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 1 month of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD8+ (<0.200x103/MicroL at month 1)) and graft survival throughout the first year of evolution.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 1 month of transplantation on the incidence of acute rejection throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 1 month of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD8+ (<0.200x103/MicroL at month 1)) and the incidence of acute rejection throughout the first year of evolution.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 1 month of transplantation on vascular disease throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 1 month of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD8+ (<0.200x103/MicroL at month 1)) and vascular disease throughout the first year of evolution.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 1 month of transplantation on diabetes throughout the first year of evolution throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 1 month of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD8+ (<0.200x103/MicroL at month 1)) and diabetes throughout the first year of evolution throughout the first.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 6 months of transplantation on overall survival throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 6 months of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD3+ (<0.500x103 MicroL at 6 months)) and overall survival throughout the first year of evolution.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 6 months of transplantation on graft survival throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 6 months of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD3+ (<0.500x103 MicroL at 6 months)) and graft survival throughout the first year of evolution.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 6 months of transplantation on the incidence of acute rejection throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 6 months of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD3+ (<0.500x103 MicroL at 6 months)) and the incidence of acute rejection throughout the first year of evolution.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 6 months of transplantation on vascular disease throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 6 months of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD3+ (<0.500x103 MicroL at 6 months)) and vascular disease throughout the first year of evolution.
To analyze the influence of the renal transplant recipient's SIMPLICITY Score at 6 months of transplantation on diabetes throughout the first year of evolution throughout the first year of evolution. | Up to 12 moths from transplant
  SIMPLICITY Score at 6 months of transplantation (from 0 to 3, assigning one point to each of the following parameters: IgG hypogammaglobulinemia (<700 mg/ dL) , C3 hypocomplementemia (<83 mg/dL) and low counts in Peripheral blood of lymphocyte T CD3+ (<0.500x103 MicroL at 6 months)) and diabetes throughout the first year of evolution throughout the first.

CONTACTS AND LOCATIONS:
Overall Officials: José María Aguado, MD, Study Chair — Hospital Universitario 12 de Octubre; Daniel Serón, MD, Study Chair — Hospital Universitario Vall d´Hebrón; Ángel Alonso, MD, Study Chair — Hospital Universitario de A Coruña; Domingo Hernández Marrero, MD, Principal Investigator — Hospital Carlos Haya; Álex Gutiérrez Dalmau, MD, Principal Investigator — Hospital Miguel Servet; Roberto Gallego, MD, Principal Investigator — Hospital Dr. Negrín; Juan Carlos Ruiz, MD, Principal Investigator — Hospital Marqués de Valdecilla; Frederic Cofàn, MD, Principal Investigator — Hospital Clinic of Barcelona; José M Cruzado, MD, Principal Investigator — Hospital Universitari de Bellvitge; Daniel Serón, MD, Principal Investigator — Hospital Universitario Vall d´Hebrón; María José Pérez Sáez, MD, Principal Investigator — Hospital del Mar; Miguel Angel Muñoz Cepeda, MD, Principal Investigator — Hospital Virgen de la Salud; Ángel Alonso, MD, Principal Investigator — Hospital Universitario de A Coruña; Gonzalo Gómez, MD, Principal Investigator — Hospital Son Espases; Amado Andrés, MD, Principal Investigator — Hospital Universitario 12 de Octubre; José Mª Portolés, MD, Principal Investigator — Hospital Universitario Puerta de Hierro Majadahonda; Roberto Marcén, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Luisa Jimeno Garcia, MD, Principal Investigator — Hospital Virgen de la Arrixaca; Luis M Pallardó Mateu, MD, Principal Investigator — Hospital Dr. Peset
Locations (15):
- Spain (15):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Vall d´Hebrón, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria, La Palmas
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 Octubre, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Carlos Haya, Málaga, Málaga
  - Hospital Virgen de la Salud, Toledo, Toledo
  - Hospital Universitario Doctor Peset, Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No